CLINICAL TRIAL: NCT03250273
Title: A Phase 2 Clinical Trial of Entinostat in Combination With Nivolumab for Patients With Previously Treated Unresectable or Metastatic Cholangiocarcinoma and Pancreatic Adenocarcinoma
Brief Title: A Clinical Trial of Entinostat in Combination With Nivolumab for Patients With Previously Treated Unresectable or Metastatic Cholangiocarcinoma and Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Syndax Pharmaceuticals (Industry); Bristol-Myers Squibb (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1798; IRB00142149 (Other: JHMI IRB); 5P01CA247886 (NIH)
Record Dates: First submitted 2017-07-28; First posted 2017-08-15 (Actual); Results first posted 2021-12-16 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Cholangiocarcinoma; Cholangiocarcinoma; Pancreatic Cancer; Metastatic Pancreatic Cancer; Unresectable Pancreatic Cancer; Unresectable Cholangiocarcinoma
Keywords: Immunotherapy; Nivolumab; Entinostat; Pancreatic Adenocarcinoma; Cholangiocarcinoma; Unresectable; Metastatic; PD-1; Antibody
MeSH Terms: conditions — Cholangiocarcinoma; Pancreatic Neoplasms; Neoplasm Metastasis | interventions — entinostat; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A - Cholangiocarcinoma (Experimental)
  Interventions: Drug: Entinostat; Drug: Nivolumab
- ARM B - Pancreatic Cancer (Experimental)
  Interventions: Drug: Entinostat; Drug: Nivolumab

INTERVENTIONS:
Drug: Entinostat — Entinostat (5mg) will be administered starting with 2 lead-in doses at 14 and 7 days before the first dose of nivolumab in combination with entinostat. After the lead-in dose, entinostat will be administered once a week (days 1, 8, 15, and 21 of each treatment cycle).
  Other Names: SNDX-275
  Arms: Arm A - Cholangiocarcinoma
Drug: Nivolumab — After both lead-in doses of entinostat, nivolumab (240 mg) will be administered every 2 weeks (day 1 and day 15 of a cycle).
  Other Names: OPDIVO, BMS-936558, MDX1106, ONO-4538
  Arms: Arm A - Cholangiocarcinoma
Drug: Entinostat — Entinostat (5mg) will be administered starting with 2 lead-in doses at 14 and 7 days before the first dose of nivolumab in combination with entinostat. After the lead-in dose, entinostat will be administered once a week (days 1, 8, 15, and 21 of each treatment cycle).
  Other Names: SNDX-275
  Arms: ARM B - Pancreatic Cancer
Drug: Nivolumab — After both lead-in doses of entinostat, nivolumab (240 mg) will be administered every 2 weeks (day 1 and day 15 of a cycle).
  Other Names: OPDIVO, BMS-936558, MDX1106, ONO-4538
  Arms: ARM B - Pancreatic Cancer

SUMMARY:
The proposed study is an open-label, two-arm study of entinostat plus nivolumab in patients with unresectable or metastatic cholangiocarcinoma (CCA) or pancreatic ductal adenocarcinoma (PDAC).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Have histologically or cytologically proven cholangiocarcinoma or adenocarcinoma of the pancreas that is metastatic or unresectable.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
4. Life expectancy of greater than 12 weeks.
5. Patients must have adequate organ and marrow function defined by study-specified laboratory tests.
6. Woman of child bearing potential must have a negative pregnancy test.
7. Must have progressive measurable disease.
8. Must have an accessible non-bone tumor that can be biopsied.
9. Must use acceptable form of birth control while on study.
10. Willing to provide tissue and blood samples.
11. Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

1. Chemotherapy, radiotherapy, investigational therapy, or surgery less than 3 weeks prior to trial registration
2. Prior treatment with epigenetic therapy (such as entinostat, panobinostat, vorinostat, romidepsin, 5-azacitidine, or decitabine)
3. Prior treatment with immunotherapy agents (including, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA4, etc.).
4. Hypersensitivity reaction to any monoclonal antibody.
5. History of any autoimmune disease: inflammatory bowel disease, (including ulcerative colitis and Crohn's Disease), rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus (SLE) autoimmune vasculitis (e.g., Wegener's Granulomatosis), central nervous system (CNS) or motor neuropathy considered to be of autoimmune origin (e.g., Guillain-Barre Syndrome, Myasthenia Gravis, Multiple Sclerosis). Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event).
6. Have significant and/or malignant pleural effusion
7. Has a pulse oximetry < 92% on room air.
8. Known history or evidence of brain metastases.
9. Conditions, including alcohol or drug dependence, intercurrent illness, or lack of sufficient peripheral venous access, that would affect the patient's ability to comply with study visits and procedures.
10. Are pregnant or breastfeeding.
11. Infection with HIV or hepatitis B or C.
12. Patients on immunosuppressive agents.
13. Requiring concurrent administration of valproic acid.
14. Patients with diverticulitis, intra-abdominal abscess, or GI obstruction
15. Any contraindication to oral agents.
16. Another active malignancy ≤ 3 years prior to registration with the exception of non-melanotic skin cancer or carcinoma-in-situ of any type.
17. Unwilling or unable to follow the study schedule for any reason.
18. Evidence of ascites on imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nilofer Azad, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Baretti M, Danilova L, Durham JN, Betts CB, Cope L, Sidiropoulos DN, Tandurella JA, Charmsaz S, Gross N, Hernandez A, Ho WJ, Thoburn C, Walker R, Leatherman J, Mitchell S, Christmas B, Saeed A, Gaykalova DA, Yegnasubramanian S, Fertig EJ, Coussens LM, Yarchoan M, Jaffee E, Azad NS. Entinostat in combination with nivolumab in metastatic pancreatic ductal adenocarcinoma: a phase 2 clinical trial. Nat Commun. 2024 Nov 12;15(1):9801. doi: 10.1038/s41467-024-52528-7. PMID 39532835

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 enrolled participant withdrew consent prior to initiating treatment
Period: Overall Study
Arm/Group | Arm A - Cholangiocarcinoma | ARM B - Pancreatic Cancer
Started | 13 | 30
Completed | 11 | 18
Not Completed | 2 | 12
Not completed — Disease Progression | 2 | 11
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - Cholangiocarcinoma | ARM B - Pancreatic Cancer | Total
Number analyzed (Participants) | 13 | 30 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 16 | 26
  >=65 years | 3 | 14 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 13 | 17
  Male | 9 | 17 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 11 | 27 | 38
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 12 | 28 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 30 | 43

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Using Response Evaluation Criteria for Solid Tumors (RECIST 1.1)
Description: Objective Response Rate (ORR) is defined as the number of patients achieving a complete response (CR) or partial response (PR) based on RECIST 1.1 criteria. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions. Subjects who discontinue due to clinical progression prior to post-baseline tumor assessments were considered as non-responders.
Time Frame: 27 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Cholangiocarcinoma | ARM B - Pancreatic Cancer
Number analyzed (Participants) | 13 | 27
Participants | 0 | 3

2. Secondary Outcome: Number of Patients Experiencing a Grade 3 or Above Treatment-related Adverse Event (AE)
Description: When calculating the incidence of AEs, each AE (as defined by NCI CTCAE v4.03) will be counted only once for a given subject.
Time Frame: 29 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Cholangiocarcinoma | ARM B - Pancreatic Cancer
Number analyzed (Participants) | 13 | 30
Participants | 5 | 19

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the duration of time from start of study treatment to time of death (OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis). Estimation based on the Kaplan-Meier curve.
Time Frame: 38 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A - Cholangiocarcinoma | ARM B - Pancreatic Cancer
Number analyzed (Participants) | 13 | 30
months | 6.378 [3.748 to NA] — Upper bound confidence interval was not reached. | 2.729 [1.84 to 5.62]

4. Secondary Outcome: Overall Survival (OS) at 6 Months
Description: OS is defined as the proportion of subjects who are alive at 6 months. Estimation based on the Kaplan-Meier curve.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A - Cholangiocarcinoma | ARM B - Pancreatic Cancer
Number analyzed (Participants) | 13 | 30
proportion of participants | 0.538 [0.326 to 0.891] | 0.277 [0.153 to 0.498]

5. Secondary Outcome: Overall Survival (OS) at 12 Months
Description: OS is defined as the proportion of subjects who are alive at 12 months. Estimation based on the Kaplan-Meier curve.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A - Cholangiocarcinoma | ARM B - Pancreatic Cancer
Number analyzed (Participants) | 13 | 30
proportion of participants | 0.308 [0.136 to 0.695] | 0.138 [0.056 to 0.343]

6. Secondary Outcome: Overall Survival (OS) at 24 Months
Description: OS is defined as the proportion of subjects who are alive at 24 months. Estimation based on the Kaplan-Meier curve.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A - Cholangiocarcinoma | ARM B - Pancreatic Cancer
Number analyzed (Participants) | 13 | 30
proportion of participants | 0.077 [0.012 to 0.506] | 0.035 [0.005 to 0.237]

7. Secondary Outcome: Overall Survival (OS) at 36 Months
Description: OS is defined as the proportion of subjects who are alive at 36 months. Estimation based on the Kaplan-Meier curve.
Time Frame: 36 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A - Cholangiocarcinoma | ARM B - Pancreatic Cancer
Number analyzed (Participants) | 13 | 30
proportion of participants | 0.077 [0.012 to 0.506] | 0.035 [0.005 to 0.237]

8. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response (DOR) will be calculated for subjects who achieve a best overall response of CR or PR. DOR is defined as the number of months from the start date of PR or CR (whichever response is recorded first) and subsequently confirmed to the first date that recurrent or progressive disease or death is documented. Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions.
Time Frame: 27 months
Population: There were no responses (PR or CR) observed in Arm A; therefore, the number of analyzed participants is zero. 3 participants achieved response in Arm B.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A - Cholangiocarcinoma | ARM B - Pancreatic Cancer
Number analyzed (Participants) | 0 | 3
months |  | 10.2 [3.7 to 17.9]

9. Secondary Outcome: Progression Free Survival (PFS) at 6 Months
Description: PFS is defined as the proportion of patients without disease progression (PD or relapse from CR) or death due to any cause at 6 months. Disease progression will be assessed using RECIST (version 1.1). Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions, Stable Disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.Estimation based on the Kaplan-Meier curve.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A - Cholangiocarcinoma | ARM B - Pancreatic Cancer
Number analyzed (Participants) | 13 | 30
proportion of participants | 0 [NA to NA] — All patients progressed by 6 months | 0.067 [0.017 to 0.254]

10. Secondary Outcome: Progression Free Survival (PFS) at 12 Months
Description: PFS is defined as the proportion of patients without disease progression (PD or relapse from CR) or death due to any cause at 12 months. Disease progression will be assessed using RECIST (version 1.1). Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions, Stable Disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.Estimation based on the Kaplan-Meier curve.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A - Cholangiocarcinoma | ARM B - Pancreatic Cancer
Number analyzed (Participants) | 13 | 30
proportion of participants | 0 [NA to NA] — All patients progressed by 12 months. | 0.067 [0.017 to 0.254]

11. Secondary Outcome: Progression Free Survival (PFS) at 24 Months
Description: PFS is defined as the proportion of patients without disease progression (PD or relapse from CR) or death due to any cause at 24 months. Disease progression will be assessed using RECIST (version 1.1). Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions, Stable Disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.Estimation based on the Kaplan-Meier curve.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A - Cholangiocarcinoma | ARM B - Pancreatic Cancer
Number analyzed (Participants) | 13 | 30
proportion of participants | 0 [NA to NA] — All patients progressed by 24 months | 0 [NA to NA] — All patients progressed by 24 months

ADVERSE EVENTS:
Time Frame: 29 months
Description: Adverse reporting collection was conducted by regular investigator assessment and laboratory measurements.
Arm/Group | Arm A - Cholangiocarcinoma | ARM B - Pancreatic Cancer
All-Cause Mortality (participants affected / at risk) | 0/13 | 1/30
Serious Adverse Events (participants affected / at risk) | 4/13 | 3/30
Other Adverse Events (participants affected / at risk) | 12/13 | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Cholangiocarcinoma (N=13) | ARM B - Pancreatic Cancer (N=30)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0)
Pneumonitis (Infections and infestations) | 2 (2) | 0 (0)
Transaminitis (Investigations) | 1 (1) | 0 (0)
Renal tubular acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Cholangiocarcinoma (N=13) | ARM B - Pancreatic Cancer (N=30)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 9 (14)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (4)
Dry lips (Gastrointestinal disorders) | 1 (1) | 0 (0)
Early satiety (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 4 (5)
Nausea (Gastrointestinal disorders) | 6 (8) | 10 (11)
Vomiting (Gastrointestinal disorders) | 0 (0) | 6 (7)
Chills (General disorders) | 0 (0) | 2 (3)
Edema (General disorders) | 4 (4) | 4 (4)
Fatigue (General disorders) | 12 (18) | 20 (25)
Fever (General disorders) | 1 (1) | 3 (7)
Flu-like symptoms (General disorders) | 1 (1) | 0 (0)
Thrush (Infections and infestations) | 2 (2) | 4 (4)
Lymphocyte count decreased (Investigations) | 2 (2) | 8 (15)
Neutrophil count decreased (Investigations) | 1 (1) | 4 (6)
Platelet count decreased (Investigations) | 3 (8) | 3 (4)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 5 (6) | 15 (17)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 3 (6)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Weight loss (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 2 (4)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (7) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4) | 4 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/73/NCT03250273/Prot_SAP_000.pdf